CLINICAL TRIAL: NCT00599170
Title: Rituximab Plus CHOP Given Every Two Weeks With Sargramostim in Patients With Newly Diagnosed Diffuse Large B-Cell Lymphoma
Brief Title: Rituximab Plus CHOP With Sargramostim in Patients With Newly Diagnosed Diffuse Large B-Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13nhl-07-3
Record Dates: First submitted 2008-01-11; First posted 2008-01-23 (Estimated); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Diffuse, Large B-Cell, Lymphoma
Keywords: This is a standard phase II trial, in which patients with newly diagnosed diffuse large B cell lymphoma will receive R-CHOP with GM-CSF
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1 (Experimental): Rituximab 375 mg/m2 iv on day 1 q 15 days just prior to CHOP, beginning with cycle 1.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — 375 mg/m2 IV

SUMMARY:
The use of R-CHOP, given every two weeks, will be associated with improvements in response rate, and progression-free survival, when compared to R-CHOP given every three weeks. The addition of sargramostim will allow safer adminIstration of the dose-intensified R-CHOP, while at the same time, improving the functional capability of the macrophages, and thus increasing the likelihood of improved clinical response and disease-free survival.

The current phase II study is being proposed in order to develop preliminary data on the efficacy and toxicity of this approach, for future study in larger, phase III randomized trials. Laboratory correlates of response will also be studied, including activation markers on monocytes/macrophages before and after sargramostim exposure; and presence or absence of informative Fc gamma III polymorphisms.

ELIGIBILITY:
Inclusion Criteria:

1. Previously untreated, histologically or cytologically documented diffuse large B cell non-Hodgkin's lymphoma.
2. Lymphoma must be CD20 positive.
3. All stages of disease.
4. Measurable or non-measurable tumor parameter(s). Non-measurable tumor parameters will be defined as not having bi-dimensional measurements (i.e. gastric or marrow involvement) but can be followed for response by other diagnostic tests such as gallium, PET imaging and/or bone marrow biopsy.
5. Age ≥ 18 years.
6. KPS ≥ 50% (ECOG PS 0, 1, or 2).
7. Able to give signed informed consent.
8. Adequate hepatic function: bilirubin ≤ 2.0 mg/dl (unless elevated secondary to lymphomatous involvement of liver or biliary system. For bilirubin > 3.0 due to hepatic involvement, the initial dose of doxorubicin will be decreased by 50%, and the initial dose of vincristine will be omitted. SGOT <5X upper limit of normal.
9. Adequate renal function: creatinine < 2.0 mg/dl, or creatinine clearance ≥ 60 ml/min, unless secondary to renal involvement by lymphoma.
10. Adequate hematologic function: granulocytes (ANC) >1000/mm3, platelets > 75,000/dl, unless these parameters are abnormal secondary to lymphomatous involvement of bone marrow. All patients must be off colony stimulating factor therapy at least 24 hours prior to institution of cycle #1 chemotherapy.
11. Left ventricular ejection fraction that is at or above the lower institutional limits of normal, as assessed by nuclear scan or echocardiogram obtained within 6 weeks of registration.
12. Concurrent radiation with or without steroids for emergency conditions secondary to lymphoma (i.e. CNS tumor, cord compression, etc) will be permitted, provided that additional, measurable or evaluable sites of lymphomatous disease are present at study entry.
13. Female patients must have a negative pregnancy test within 72 hours of entering into the study. Both men and women will be included and, if of child bearing potential, must agree to use adequate contraception for the duration of the treatment. Women must avoid pregnancy and men avoid fathering children while in the study.

    -

Exclusion Criteria:

1. Presence of second active tumor, other than non melanomatous skin cancer, carcinoma in situ of the cervix.
2. Primary central nervous system lymphoma, including parenchymal brain or spinal cord lymphoma.
3. Pregnant women or nursing mothers.
4. ECOG performance score 3 or more (KPS <50%).
5. Expected survival < 3 months.
6. Unable to comply with the requirements of the protocol, or unable to provide adequate informed consent in the opinion of the principal investigator.
7. Serious, on-going non-malignant disease or infection, which, in the opinion of the investigator and/or the sponsor, would compromise other protocol objectives.
8. Major surgery, other than diagnostic surgery, within four weeks.
9. History of prior therapy with Rituximab within 12 months. Patients treated with Rituximab more than 12 months earlier are eligible only if it was given for indications other than the treatment of aggressive lymphoma.
10. History of prior cytotoxic chemotherapy or radiotherapy for this lymphoma.
11. History of cutaneous or muco-cutaneous reactions or diseases in the past, due to any cause, severe enough to cause hospitalization or an inability to eat or drink for 2 days or more. This exclusion relates to the long-term possibility of severe muco-cutaneous or cutaneous reactions to Rituximab, which maybe occurred at increased frequency in patients who have had severe skin disease or reactions in the past.
12. Any acute inter-current infection that may interfere with planned protocol treatment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2008-01-10 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2021-01-10 (Actual)

PRIMARY OUTCOMES:
The primary endpoint in this trial will be tumor complete response (CR, CRu) to R-CHOP + GM-CSF, given every 14 days | Every 2 cycles

SECONDARY OUTCOMES:
Response duration | Every 2 cycles

CONTACTS AND LOCATIONS:
Overall Officials: Anil Tulpule, MD, Principal Investigator — University of Southern California
Locations (1):
- USC Norris Comprehensive Cancer Center, Los Angeles, California, United States